CLINICAL TRIAL: NCT01498835
Title: Phase 1 Trial of Concurrent Sunitinib and Radiation Therapy as Preoperative Treatment for Locally Advanced or Recurrent Soft Tissue Sarcoma.
Brief Title: Safety Study of Preoperative Sunitinib and Radiation in Soft Tissue Sarcoma
Acronym: SunRaSe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Peter Hohenberger, MD PhD, Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GISG 03; 2007-002864-87 (EudraCT Number)
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Soft Tissue Sarcoma
Keywords: Soft tissue sarcoma; Radiation therapy; Sunitinib
MeSH Terms: conditions — Sarcoma | interventions — Sunitinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Combined Sunitinib and irradiation (Experimental): Patients with locally advanced or recurrent soft tissue sarcoma will receive Sunitinib and irradiation as neoadjuvant treatment. Restaging and tumor resection will be performed 6 weeks after completion of sunitinib and irradiation.
  Interventions: Drug: Sunitinib

INTERVENTIONS:
Drug: Sunitinib — Patients will receive Sunitinib daily for 2 weeks prior to and then concurrently with irradiation as neoadjuvant treatment. Radiotherapy will be given as intensity modulated radiation therapy with a total dose of 50.4Gy in 28 fractions to each patient (5 1/2 weeks).
  Sunitinib will be given in two dose levels. The first dose level will be 25mg Sunitinib per os daily. The second dose level will be 37.5mg sunitinib per os daily. A dose modification schedule according to a 3+3 design will be applied for patient accrual.
  Other Names: Radiation therapy

SUMMARY:
To evaluate the toxicity of sunitinib concurrently given with irradiation for preoperative treatment of locally advanced or recurrent soft tissue sarcoma.

DETAILED DESCRIPTION:
Although the introduction of multimodal treatment of soft tissue sarcoma resulted in great progress in STS treatment, local failure still occurs in 10-20% of STS patients. Therefore further improvement of local and systemic treatment is needed in order to achieve tumor control and limb salvage. The proposed study treatment will combine external beam radiation and orally administered sunitinib.

Sunitinib is a multiple receptor tyrosine kinase (RTK) inhibitor with anti-angiogenic and anti-tumoral properties. For their key role in tumor development, RTKs are regarded as excellent targets for cancer chemotherapy. External beam radiation is widely used as neoadjuvant treatment for locally advanced soft tissue sarcoma.

The concurrent application of anti-angiogenic sunitinib appears reasonable, since STS are highly vascularized tumors and overexpression of VEGFR and other RTKs has been shown for various histologic soft tissue sarcoma subtypes. At first sight, the combination of antiangiogenic treatment and radiation seems to be contradictory, since anti-angiogenic treatment attacks tumor vasculature and radiation effects are decreased by hypoxia. Yet, in animal studies the concurrent application of radiation with tyrosine kinase inhibitors such as sunitinib or other antiangiogenic agents resulted in additive, if not synergistic antitumoral effects. These results can be explained by the superiority of the anti-tumoral activity of antiangiogenic agents over their hypoxia related, radiation weakening effects; or by the hypothesis of vascular normalization. It is well known that tumor vasculature is immature and ineffective in means of blood supply and oxygenation. In preclinical models, antiangiogenic agents balanced pro- and anti-angiogenic effectors which may result in maturation of tumor vasculature with improvement of blood flow and oxygen supply.

The combination of sunitinib as an anti-angiogenic and anti-proliferative agent thus might not only add the therapeutic effects of the RTK-inhibitor and external beam radiation but might additionally lead to a radiosensitizing effect due to tumor vessel normalization. The Purpose of this study is to assess the toxicity of the combined treatment and to gather preliminary data on treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven soft tissue sarcoma of any histology but GIST, Angiosarcoma, dermatofibrosarcoma protuberans, Ewing Sarcoma or Embryonal Rhabdomyosarcoma
* patients with primary tumors OR with local recurrences who did not receive prior radiation therapy OR with solitary metastatic lesions may be included
* complete resection after neoadjuvant treatment is expected
* age of 18 or older
* ECOG performance score 0 or 1
* normal organ and bone marrow function
* ability to give written informed consent

Exclusion Criteria:

* medication with inhibitors or inducers of CYP3A4
* prior therapy with tyrosine kinase inhibitors or conventional chemotherapy within 4 weeks before study inclusion
* history of myocardial infarction, stroke or thromboembolic events
* clinical signs of heart failure (NYHA 3 or 4)
* anticoagulation with Vitamin K antagonists
* acquired or hereditary coagulopathy
* uncontrolled hypertension
* uncontrolled intercurrent illness
* women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-02; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the dose limiting toxicity and maximal tolerated dose of sunitinib given concurrently with irradiation as neoadjuvant treatment in soft tissue sarcoma. | 12 weeks
  Toxicity of the study treatment will be documented according to CTCAE 4.0 during and until 4 weeks after study treatment.

SECONDARY OUTCOMES:
To evaluate the response to sunitinib given concurrently with radiation as neoadjuvant treatment in soft tissue sarcoma. | 6 weeks after completion of study treatment.
  Imaging response will be determined according to RECIST criteria comparing magnetic resonance imaging performed prior to and 6 weeks after completion of study treatment. Pathologic response will be determined evaluating the the fraction of non-viable tumor in the resection specimen.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hohenberger, MD PhD, Principal Investigator — Heidelberg University
Locations (2):
- Germany (2):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - University Medical Center Mannheim, Mannheim

REFERENCES:
- [Derived] Jakob J, Simeonova A, Kasper B, Ronellenfitsch U, Rauch G, Wenz F, Hohenberger P. Combined sunitinib and radiation therapy for preoperative treatment of soft tissue sarcoma: results of a phase I trial of the German interdisciplinary sarcoma group (GISG-03). Radiat Oncol. 2016 Jun 3;11:77. doi: 10.1186/s13014-016-0654-2. PMID 27255678
- [Derived] Jakob J, Rauch G, Wenz F, Hohenberger P. Phase I trial of concurrent sunitinib and radiation therapy as preoperative treatment for soft tissue sarcoma. BMJ Open. 2013 Sep 18;3(9):e003626. doi: 10.1136/bmjopen-2013-003626. PMID 24048627